CLINICAL TRIAL: NCT01763853
Title: Impact of Fluid Resuscitation Therapy on Pulmonary Edema as Measured by Alveolar Fluid Clearance in Patients With Acute Respiratory Distress Syndrome (ARDS)
Acronym: IROCA
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Clermont-Ferrand (Other)
Collaborators: R2D2 Retinoids, Reproduction Developmental Diseases (Other); Université d'Auvergne (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CHU-0134
Record Dates: First submitted 2012-12-10; First posted 2013-01-09 (Estimated); Last update posted 2016-07-29 (Estimated); Status verified 2016-07

CONDITIONS: Acute Respiratory Distress Syndrome (ARDS); Hypovolemia; Pulmonary Edema
Keywords: Acute respiratory distress syndrome (ARDS); Pulmonary edema; Alveolar fluid clearance; Alveolar epithelial dysfunction; Receptor for advanced glycation end-products (RAGE); Fluid resuscitation therapy; Hypovolemia; Crystalloid; Hydroxyethyl Starch; Intensive care unit
MeSH Terms: conditions — Respiratory Distress Syndrome; Hypovolemia; Pulmonary Edema | interventions — Albumins

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- albumin (Other): The main objective of our prospective double blind, randomized, controlled trial is to compare the rate of alveolar fluid clearance, a marker of alveolar edema fluid resorption, in 2 groups of patients with ARDS and suffering from hypovolemia: those treated with albumin and those treated with crystalloid (fluid challenge of 7 mL/kg over 15 minutes, that can be repeated 3 times if hypovolemia persists).
  Interventions: Drug: 4% albumin
- crystalloid (Other): The main objective of our prospective double blind, randomized, controlled trial is to compare the rate of alveolar fluid clearance, a marker of alveolar edema fluid resorption, in 2 groups of patients with ARDS and suffering from hypovolemia: those treated with albumin and those treated with crystalloid (fluid challenge of 7 mL/kg over 15 minutes, that can be repeated 3 times if hypovolemia persists).
  Interventions: Drug: 4% albumin

INTERVENTIONS:
Drug: 4% albumin

SUMMARY:
The need for fluid resuscitation (FR) in ICU patients with acute respiratory distress syndrome (ARDS) is common. Indeed, relative or absolute hypovolemia is a common phenomenon that the intensivist must recognize early and treat promptly. Fluid challenge may have adverse side effects associated with fluid administration. The diffusion within the interstitial space may favor edema formation and cause cardiac dysfunction by volume overload. Edema formation is global and may specifically alter pulmonary alveolar epithelial integrity, leading to enhanced alveolar edema and impaired gas exchange.

Currently, two types of fluids are frequently used, crystalloids and colloids. Among colloids and compared to crystalloids, albumin has the theoretical advantage of causing greater volume expansion.

We hypothesized that a fluid resuscitation therapy with albumin generates less pulmonary edema than a fluid resuscitation therapy with crystalloids.

The aim of our study is to compare alveolar fluid clearance, as a marker of alveolar edema fluid resorption, in 2 groups of patients: those treated with albumin and those treated with crystalloid.

DETAILED DESCRIPTION:
The main objective of our prospective double blind, randomized, controlled trial is to compare the rate of alveolar fluid clearance, a marker of alveolar edema fluid resorption, in 2 groups of patients with ARDS and suffering from hypovolemia: those treated with albumin and those treated with crystalloid (fluid challenge of 7 mL/kg over 15 minutes, that can be repeated 3 times if hypovolemia persists).

The evolution of respiratory and hemodynamic parameters, as measured by transpulmonary thermodilution (extra-vascular lung water, pulmonary vascular permeability index, cardiac output, global enddiastolic volume), plasma osmolality, plasma oncotic pressure and plasma levels of brain natriuretic peptid (BNP) will be studied one hour and 3 hours after after fluid resuscitation in the two groups. In order to evaluate alveolar epithelial dysfunction in patients receiving either albumin or crystalloid, plasma and alveolar levels of sRAGE (the soluble form of the receptor for advanced glycation endproducts) will be measured by ELISA. Lung aeration and fluid-induced derecruitment will be evaluated with an electrical impedance tomograph (PulmoVista®500, Dräger).

ELIGIBILITY:
Inclusion Criteria:

* ICU patients under mechanical ventilation
* Patients within the first 24 hours after onset of moderate or severe ARDS, as defined by the Berlin definition (JAMA. 2012;307(23):2526-2533)
* Hypovolemia requiring fluid resuscitation therapy

Exclusion Criteria:

* Pregnancy
* Age under 18
* Refusal of the protocol
* Contraindications for the use of Voluven© or Ringer Lactate©
* Contraindications for femoral artery catheterization or subclavian venous catheterization

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2012-12; Primary Completion 2017-04 (Estimated); Study Completion 2017-05 (Estimated)

PRIMARY OUTCOMES:
Rate of alveolar fluid clearance | one hour after administration of fluid resuscitation

SECONDARY OUTCOMES:
Extra-vascular lung water | one hour and three hours after administration of fluid resuscitation
Pulmonary vascular permeability index | one hour and three hours after administration of fluid resuscitation
Global enddiastolic volume index | one hour and three hours after administration of fluid resuscitation
mean arterial pressure | one hour and three hours after administration of fluid resuscitation
cardiac output | one hour and three hours after administration of fluid resuscitation
pulse pressure variation | one hour and three hours after administration of fluid resuscitation
stroke volume variation | one hour and three hours after administration of fluid resuscitation
central venous venous oxygenation | one hour and three hours after administration of fluid resuscitation
central venous pressure | one hour and three hours after administration of fluid resuscitation
PaO2 | one hour and three hours after administration of fluid resuscitation
lung compliance | one hour and three hours after administration of fluid resuscitation
airways resistance | one hour and three hours after administration of fluid resuscitation
lung injury score | one hour and three hours after administration of fluid resuscitation
Plasma levels of sRAGE | one hour and three hours after administration of fluid resuscitation
Alveolar levels of sRAGE | one hour and three hours after administration of fluid resuscitation
Brain natriuretic peptide levels | one hour and three hours after administration of fluid resuscitation
Plasma osmolarity | one hour and three hours after administration of fluid resuscitation
Oncotic pressure | one hour and three hours after administration of fluid resuscitation
Electrical impedance tomography | one hour and three hours after administration of fluid resuscitation
Mortality | Day 20, Day 90

CONTACTS AND LOCATIONS:
Overall Officials: Matthieu JABAUDON, Principal Investigator — University Hospital, Clermont-Ferrand
Locations (1):
- CHU Clermont-Ferrand, Clermont-Ferrand, France